CLINICAL TRIAL: NCT06456411
Title: Real-Time Evaluation of Severity of Perceived Pain in Patients With Cancer by Using Functional Near-Infrared Spectroscopy (fNIRS), and Investigation of Pain Relief Utilizing Virtual Reality Technologies
Brief Title: Functional Near-Infrared Spectroscopy and Virtual Reality Relaxation Programs for Pain Management in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: I 1720121; NCI-2021-11854 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 1720121 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma; Kidney Carcinoma; Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Renal Cell; Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A (fNIRS) (Experimental): Participants undergo fNIRS for 10 minutes.
  Interventions: Procedure: Functional Near-Infrared Spectroscopy; Other: Questionnaire Administration
- Group B (fNIRS, VR) (Experimental): Patients undergo fNIRS for 10 minutes followed by a relaxation period using VR for over 15 minutes.
  Interventions: Procedure: Functional Near-Infrared Spectroscopy; Other: Questionnaire Administration; Other: Virtual Technology Intervention
- Group C (fNIRS) (Experimental): Patients undergo fNIRS for 10 minutes.
  Interventions: Procedure: Functional Near-Infrared Spectroscopy; Other: Questionnaire Administration
- Group D Arm 1 - VR (Experimental): Patients undergo Therapeutic VR program for up to 30 minutes four times per week
  Interventions: Other: Virtual Technology Intervention
- Group D Arm II - Sham VR (Experimental): Patients undergo placebo VR program for up to 30 minutes four times per week.
  Interventions: Other: Virtual Technology Intervention
- Group E (Experimental): Cold stimulation on day 1 of each chemotherapy cycle and day 3.
  Interventions: Other: Cold Stimulation

INTERVENTIONS:
Procedure: Functional Near-Infrared Spectroscopy — Undergo fNIRS
  Other Names: fNIRS; Functional Near Infrared Spectroscopy; Functional NIR Spectroscopy; Functional Optical Brain Imaging
  Arms: Group A (fNIRS); Group B (fNIRS, VR); Group C (fNIRS)
Other: Questionnaire Administration — Ancillary studies
  Arms: Group A (fNIRS); Group B (fNIRS, VR); Group C (fNIRS)
Other: Virtual Technology Intervention — Undergo relaxation period using VR
  Other Names: Virtual Reality Intervention; Virtual Technology
  Arms: Group B (fNIRS, VR); Group D Arm 1 - VR; Group D Arm II - Sham VR
Other: Cold Stimulation — cold stimulation using ice pack
  Other Names: ice pack
  Arms: Group E

SUMMARY:
This study aims to develop objective tools for assessing perceived pain severity in cancer patients and survivors, evaluate the sustained effectiveness of non-pharmacological interventions such as virtual reality in reducing pain and medication use, and create tools for the early detection of neuropathy. Wireless, non-invasive neuroimaging methods, including functional near-infrared spectroscopy (fNIRS), will be used to support these objectives

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop an algorithm for objective evaluation of pain severity and distinguish the location of pain without needing patient cooperation.

II. Find the relationship between fNIRS (functional near-infrared spectroscopy) features and severity of pain as well as the relationship (if any) between perceived pain severity and psychological factors.

III. Understand the acute cold dysesthesias with oxaliplatin and how this correlated with more chronic neuropathy IV. Investigate the sustained effects of therapeutic virtual reality versus Sham virtual reality on pain severity and medication doses.

V. Monitor VR-induced changes of brain activity to find out the underlying mechanisms of pain alleviation.

SECONDARY OBJECTIVES:

I. Investigate the effect of demographic factors on perceived pain severity and VR-inducated pain alleviation

- Investigate the effects of repeated VR use on doses of medications.

OUTLINE: Healthy participants are assigned to group A. Cancer patients are randomized to group B, C , D or E.

GROUP A: Participants undergo fNIRS for 10 minutes.

GROUP B: Patients undergo fNIRS for 10 minutes followed by a relaxation period using virtual reality (VR) for over 15 minutes.

GROUP C: Patients undergo fNIRS for 10 minutes.

GROUP D: Patients are randomized to 1 of 2 arm:

ARM I - Patients use VR for up to 30 minutes.

ARM II: Patients use Sham VR Program for up to 30 minutes

GROUP E: Cold pack stimulation on Day 1 of each chemotherapy cycle and day 3.

ELIGIBILITY:
Inclusion Criteria: GROUPS A, B and C:

* Participants in Group A, B or C (cancer pts as well as healthy volunteers) must be over the age of 18
* Participants in Groups A or C (cancer pts as well as healthy volunteers) need to be able to be in a sedentary posture for approximately 20 minutes
* Participants in Group B and C: Patient can be in any stage of cancer treatment, such as diagnosis, treatment (surgery, chemotherapy, immunotherapy, radiation), recovery, remission and is experiencing acute pain from treatment or cancer itself. Cancers include but are not limited to: breast, thoracic, lung, kidney, colon, pancreatic, etc.
* Must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Participants in Group B and C must be free from other forms of chronic pain, e.g., rheumatologic pain, must be free from neurologic illnesses, e.g., stroke, and must have no brain metastases which could interfere with brain functions

Inclusion Criteria - GROUP D:

* Men and women of 40-80 yrs old
* Stage I-III lung cancer survivors who have undergone lung resection and developed persistent post-thoracotomy pain (PPTP)
* Willing to comply with study procedures
* Be able to remain sedentary for 20 minutes during functional near-infrared spectroscopy (fNIRS) data recording sessions, including 10 minutes each for fNIRS system setup and 10 minutes data recording.
* Must understand the investigational nature of the study and sign a written informed consent form approved by the Independent Ethics Committee/Institutional Review Board.
* Female participants must not be pregnant to participate in this study. During the third trimester, the fetus's brain is significantly developed and may interact with the mother's brain. As this study involves recording brain activity using fNIRS, it is necessary to exclude pregnant individuals to ensure the quality of the research data.
* Be able to remove any items from their scalp that might block direct contact between the fNIRS optodes and the skin. This includes, but is not limited to, wigs and hijabs.
* Must be free from other forms of chronic pain, e.g., rheumatologic pain
* Must be free from neurologic illnesses, e.g., stroke
* Had no brain metastases which could interfere with brain functions

Inclusion criteria for Group E:

* Men and women aged 18 yrs and older.
* Diagnosed with colorectal or pancreatic cancer, scheduled to receive a 14-day cycle of oxaliplatin chemotherapy (oxaliplatin plus infusional fluorouracil regimens). Limiting the study to these patients ensures a more uniform population, reducing variability related to treatment regimens.
* Participants must be free from other forms of chronic neuropathy
* Participants must be free from neurologic illnesses, e.g., stroke
* Had no brain metastases which could interfere with brain functions
* Diabetic patients will be excluded as those patients may experience different neuropathy and their reactions might skew the results.
* Participants must be willing to comply with study procedures.
* Participants must understand the investigational nature of the study and sign a written informed consent form approved by the Independent Ethics Committee/Institutional Review Board
* Participants in Groups B and C must be free from other forms of chronic pain (e.g., rheumatologic pain), must be free from neurologic illnesses (e.g., stroke), and must have no brain metastases which could interfere with brain functions

Exclusion Criteria - GROUPS A, B and C:

* Unwilling or unable to follow protocol requirements
* Currently pregnant or planning to become pregnant during the study period
* Medical condition predisposing to nausea or dizziness.
* Hypersensitivity to flashing light or motion.
* No stereoscopic vision or severe hearing impairment.
* Unwillingness or inability to follow protocol requirements.
* Individuals with impaired decision-making capacity.
* Individuals with electronic or metallic implants in the head.
* Unable to remove any items from their scalp that might block direct contact between the fNIRS optodes and the skin. This includes, but is not limited to, wigs and hijabs
* Prisoners

  * Group B: Exclusion of individuals with hypersensitivity to flashing lights or motion. Rationale: Such hypersensitivities can increase the risk of seizures or severe discomfort when exposed to common elements of VR programs, which frequently include rapid visual and motion stimuli.
* Group B: Exclusion of individuals with impaired stereoscopic vision or severe hearing impairments.

Exclusion criteria for Group D

* individuals with hypersensitivity to flashing lights or motion. Rationale: Such hypersensitivities can increase the risk of seizures or severe discomfort when exposed to common elements of VR programs, which frequently include rapid visual and motion stimuli.
* individuals with impaired stereoscopic vision or severe hearing impairments. Rationale: VR programs often involve moving objects, flashing lights, and immersive soundscapes. Participants must have sufficient vision and hearing to effectively engage with and safely navigate these environments.
* Currently pregnant or planning to become pregnant during the study period.
* Unwillingness or inability to follow protocol requirements.
* individuals with impaired decision-making capacity. Rationale: Participants must be able to provide informed consent and make decisions regarding their continued participation in the study.
* Prisoners
* Individuals with electronic or metallic implants in the head, as these implants may obstruct direct contact between the fNIRS optodes and the skin.
* Patients with medical conditions that predispose them to nausea or dizziness. Rationale: To minimize the risk of cybersickness that may be induced by VR programs.
* Patients with signs of cancer-related cachexia, specifically those with >15% unintentional weight loss over the past 6 months or a BMI <18 will be excluded to ensure safety and data integrity.
* Diabetic patients are excluded as they may experience chronic pain differently.

Exclusion Criteria for Group E

* For Group E: Individuals treated with Carboplatin, Cisplatin, taxanes, or other platinum-based therapies should be excluded. These treatments are known to cause peripheral neuropathy, and their inclusion could confound the results. To focus specifically on neuropathy caused by oxaliplatin, patients receiving other neurotoxic chemotherapy agents are excluded.
* Individuals who underwent other neuropathy-associated chemotherapy treatments will be excluded.
* Diabetic patients will be excluded as those patients may experience neuropathy differently.
* Females who are pregnant or plan to become pregnant during the study period will be excluded.
* Unwillingness or inability to follow protocol requirements.
* individuals with impaired decision-making capacity. Rationale: Participants must be able to provide informed consent and make decisions regarding their continued participation in the study.
* Individuals who are not yet adults (younger than 18 years).
* Prisoners.
* Individuals with electronic or metallic implants in the head, as these implants may obstruct direct contact between the skin and fNIRS optodes.
* Pre-existing conditions or comorbidities that could interfere with the study, such as severe neurological disorders, uncontrolled diabetes, or peripheral neuropathy unrelated to chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2030-07-12 (Estimated); Study Completion 2030-07-12 (Estimated)

PRIMARY OUTCOMES:
Gain knowledge of Brain activity during pain | Up to 16 months
  Computational neuroscience algorithms and graph theories will be used to extract informative patterns of brain activity and diagnose the stimulated brain areas associated with pain and pain severity as well as any relationships between pain severity, functional near-infrared spectroscopy (fNIRS) measures, and visual perception.

SECONDARY OUTCOMES:
Determine if utilizing virtual reality technologies significantly alleviate pain through distraction | Up to 16 months
  By utilizing virtual reality relaxation program we will analyze brain activity to find out how this distraction is controlled by the brain.
Reason for pain alleviation caused by virtual reality techniques | Up to 16 months
  Measured by fNIRS and quantified by signal processing and network neuroscience algorithms, to find out the reason for pain alleviation caused by virtual reality techniques. We will also investigate if cognitive distraction can be the main reason.

CONTACTS AND LOCATIONS:
Overall Officials: Somayeh B Shafiei, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States